CLINICAL TRIAL: NCT05199272
Title: A Phase 1/2a, Multicenter, Open-Label, Dose-Escalation and Expansion Study of Intravenously Administered 23ME-00610 in Patients With Advanced Solid Malignancies
Brief Title: A Phase 1/2a Study of 23ME-00610 in Patients With Advanced Solid Malignancies
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: 23andMe, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 23ME-00610-CLIN-001
Record Dates: First submitted 2022-01-06; First posted 2022-01-20 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-05

CONDITIONS: Solid Tumor; Clear Cell Renal Cell Carcinoma; Epithelial Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Carcinoma; Neuroendocrine Tumors; MSI-H Cancer; Cancer With A High Tumor Mutational Burden; Extensive-stage Small-cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell; Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms; Neuroendocrine Tumors; Small Cell Lung Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A (Experimental): Patients will receive escalating doses of 23ME-00610
  Interventions: Drug: 23ME-00610
- Part B (Experimental): Patients will receive the recommended dose(s) of 23ME-00610
  Interventions: Drug: 23ME-00610

INTERVENTIONS:
Drug: 23ME-00610 — 23ME-00610 given by IV infusion

SUMMARY:
This is a first-in-human open-label Phase 1/2a study to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics, and preliminary clinical activity of 23ME-00610 given by intravenous infusion in patients with advanced solid malignancies who have progressed on all available standard therapies

DETAILED DESCRIPTION:
This study includes a dose-escalation phase in Part A to determine the maximum tolerated dose (MTD) and/or recommended phase 2 dose (RP2D) followed by 6 monotherapy expansion arms in Part B to further evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics, and clinical activity of 23ME-00610 in patients with solid malignancies.

5 tumor- specific monotherapy expansion cohort will enroll up to 15 patients/cohort with the following locally advanced (unresectable) or metastatic solid malignancies:

1. Clear cell renal cell carcinoma (ccRCC)
2. Epithelial ovarian, fallopian tube or primary peritoneal carcinoma
3. Neuroendocrine cancers
4. Microsatellite instability-high (MSI-H) and/or tumor mutational burden-high (TMB-H) solid cancers and
5. Extensive stage Small cell lung cancer (ES-SCLC)

A cohort of up to 8 evaluable adolescent patients with locally advanced (unresectable), or metastatic solid cancers will also be enrolled.

Approximately 15 additional evaluable patients will be added to the cohorts with Epithelial ovarian, fallopian tube or primary peritoneal carcinoma and Neuroendocrine cancers in Part B to evaluate another dose level with pharmacologic or PD evidence of therapeutic effect below the MTD/RP2D identified in Part A (for a maximum of 30 patients in total at the alternate dose).

ELIGIBILITY:
Key Inclusion Criteria:

1. Part A: Adults ≥ 18 years of age; Part B: ≥ 12 to years of age, weighing at least 40 kg (total body weight)
2. Part A: Histologically-diagnosed locally advanced (unresectable), or metastatic solid cancer that has progressed after all available standard therapy for the specific tumor type, or for which all available standard therapy has proven to be ineffective or if no further standard therapy exists.

   Part B:
   1. Cohort 1B: Histologically-diagnosed locally advanced (unresectable) or metastatic ccRCC that has progressed following all available standard therapy (e.g., anti-PD(L)-1, anti-vascular endothelial growth factor [VEGF] kinase inhibitors), or if no further standard therapy exists.
   2. Cohort 2B: Histologically-diagnosed locally advanced (unresectable) or metastatic, platinum-resistant epithelial ovarian, fallopian tube or primary peritoneal carcinoma (i.e., disease recurrence within 6 months of completion of platinum-based therapy) that has progressed following all available standard therapy, or if no further standard therapy exists.
   3. Cohort 3B: The following histologically-diagnosed locally advanced (unresectable) or metastatic neuroendocrine cancers that have progressed following all available standard therapy, or if no further standard therapy exists:

      * Merkel cell carcinoma
      * Well-differentiated Grade 3 neuroendocrine cancers with unfavorable biology (as per National Comprehensive Cancer Network [NCCN] guidelines) from any site
      * Poorly differentiated neuroendocrine carcinoma (or extrapulmonary large and small cell carcinoma)
      * Patients with other cancers that show evidence of focal neuroendocrine differentiation may be included with approval from the medical monitor at 23andMe.
   4. Cohort 4B: Histologically-diagnosed locally advanced (unresectable) or metastatic solid cancer that has progressed following all available standard therapy, or if no further standard therapy exists and meets the following criteria:

      TMB-H solid cancer that has been confirmed by the FoundationOne CDx assay or other industry/institutional equivalent platform forTMB assessment using a cutoff of greater than or equal to 10 mutations/megabase and/or MSI-H solid cancer that has been confirmed by immunohistochemistry for MMR proteins or polymerase chain reaction (PCR) of microsatellites or MMR gene mutation by a next-generation sequencing (NGS) panel.
   5. Cohort 5B: In jurisdictions where local regulations and IRB/EC allows, adolescents with histologically-diagnosed locally advanced (unresectable), or metastatic solid cancer that has progressed after all available standard therapies for the specific tumor type, or if no further standard therapy exists.
   6. Cohort 6B: Histologically-diagnosed locally advanced (unresectable) or metastatic ES-SCLC that has progressed following all available standard therapy, or if no further standard therapy exists.
3. Part A: Adults 18+: Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1; Part B: Adolescents ≥ 12 to < 16 years of age: Lansky Play Scale ≥ 50; Adolescents ≥ 16 years of age: Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1;
4. Life expectancy ≥ 12 weeks
5. Part A: Patients without RECIST measurable disease (e.g., evaluable disease only) will be eligible for enrollment in Part A, regardless of tumor type; Part B: Patients enrolled in Part B must have measurable disease by per RECIST 1.1 and have ≥ 1 site of measurable disease that has not been previously irradiated.

Key Exclusion Criteria:

1. Females who are pregnant (positive serum pregnancy test within 7 days prior to study drug administration) or breastfeeding.
2. Immune Related Medical History:

   1. Active autoimmune disease that has required systemic disease-modifying or immunosuppressive treatment within the last 2 years
   2. Receipt of systemic immunosuppressive therapy (e.g. steroids) within 4 weeks prior to the start of study drug administration
   3. History of idiopathic pulmonary fibrosis, interstitial lung disease, organizing pneumonia, non-infectious pneumonia that required steroids, or evidence of active, non-infectious pneumonitis
   4. History of Grade ≥ 3 immune-mediated toxicity
3. Prior allogeneic or autologous bone marrow transplant, or other solid organ transplant.
4. History of a positive test for:

   1. Hepatitis C virus (HCV) infection, except for those who have completed curative therapy for HCV and have undetectable HCV RNA
   2. Hepatitis B virus (HBV) infection, except for those who are receiving treatment with HBV-active nucleos(t)ide antiviral therapy at the time of study entry and have undetectable HBV DNA
   3. Human Immunodeficiency Virus (HIV) infection, except those who meet the following criteria: CD4+ T cells ≥ 350 cells/μL, no history of Acquired Immunodeficiency Syndrome (AIDS)-defining opportunistic infections, HIV RNA < 50 copies/mL, and on a stable antiretroviral regimen for at least 3 months.
5. Prior radiation therapy with an inadequate washout between the last dose and the start of study drug, defined as follows: 1) at least 2 weeks for palliative radiation to the extremities for osseous bone metastases is required; 2) at least 4 weeks for radiation to the chest, brain, or visceral organs is required; and 3) at least 6 weeks for large-field radiation is required.
6. Prior anticancer therapy, including chemotherapy, targeted therapy, biological therapy or immune-checkpoint inhibitors within 4 weeks or 5 drug half-lives (whichever is shorter)
7. History of another malignancy in the previous 2 years, unless cured by surgery alone and continuously disease free.
8. Recent history of cardiovascular disease
9. Uncontrolled or symptomatic CNS (central nervous system) metastases and/or carcinomatous meningitis

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 141 (Estimated)
Dates: Start 2021-12-29 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Part A: Incidence and severity of dose-limiting toxicities (DLTs) | 21 days
Part B adolescents: Incidence and severity of dose-limiting toxicities (DLTs) | 21 days
Part A: Incidence and severity of adverse events (AEs) | Up to 90 days post treatment
Part B adolescents: Incidence and severity of adverse events (AEs) | Up to 90 days post treatment
Part A: Incidence and severity of serious adverse events (SAEs) | Up to 90 days post treatment
Part B adolescents: Incidence and severity of serious adverse events (SAEs) | Up to 90 days post treatment

SECONDARY OUTCOMES:
Part A: Prevalence and incidence of antidrug antibodies (ADA) to 23ME-00610 | Up to 5 days post treatment discontinuation
Overall survival (OS) | Up to 5 years

CONTACTS AND LOCATIONS:
Locations (13):
- United States (10):
  - Stanford Cancer Institute, Palo Alto, California
  - Emory University, Atlanta, Georgia
  - Karmanos Cancer Institute, Detroit, Michigan
  - R.J.Zuckerberg Cancer Center, Lake Success, New York
  - Cohen Children's Medical Center, New Hyde Park, New York
  - Oregon Health & Science University, Portland, Oregon
  - Vanderbilt University, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - START Center for Cancer Care, San Antonio, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia
- Canada (3):
  - Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - The Hospital for Sick Children, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No